CLINICAL TRIAL: NCT01849198
Title: Accelerometry at the Neck: Comparison With m. Adductor Pollicis Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kreiskrankenhaus Dormagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: NMMneck
Record Dates: First submitted 2013-04-29; First posted 2013-05-08 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Feasibility of Measurement of a Neuromuscular Block at the m. Trapezius
Keywords: accelerometry; neuromuscular block; m. trapezius

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group trapezius (Other): Assessment of intubation conditions after onset of the neuromuscular block at the m. trapezius
  Interventions: Device: accelerometry m. trapezius and m. adductor pollicis
- group adductor pollicis (Other): assessment of intubation conditions after onset of the neuromuscular block at the m. adductor pollicis
  Interventions: Device: accelerometry m. trapezius and m. adductor pollicis

INTERVENTIONS:
Device: accelerometry m. trapezius and m. adductor pollicis

SUMMARY:
Accelerometric Assessment of neuromuscular block during anaesthesia is routinely performed at the M. adductor pollicis. However, many operations require positioning of the patients with arms attached to the body. In these situations, the anaesthesiologist has no access to the m.adductor pollicis.

In this study, a new position of accelerometry at the neck is evaluated: Stimulation of the n. accessorius with accelerometry of the m. trapezius.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anaesthesia with endotracheal intubation
* weight 50-90 kg

Exclusion Criteria:

* Pregnancy
* allergy to one of the drugs used
* risk of pulmonary aspiration
* expected difficulties with endotracheal intubation
* intake of drugs known to influence neuromuscular block
* infection (CRP > 0,5 mg/dl, leukocyte count > 12000/µl)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Recovery to a train of four ratio of 0.9 | 60 minutes
  Comparison between time to recovery [s] to a train of four ratio of 0.9 between both groups

SECONDARY OUTCOMES:
onset of neuromuscular block | 10 min
  Comparison of onset time [s] between both groups. Onset time is defined as decrease of T1 to < 5% of initial twitch height.

CONTACTS AND LOCATIONS:
Locations (1):
- KKH Dormagen, Dormagen, Germany

REFERENCES:
- [Derived] Soltesz S, Stark C, Noe KG, Anapolski M, Mencke T. Comparison of the trapezius and the adductor pollicis muscle as predictor of good intubating conditions: a randomized controlled trial. BMC Anesthesiol. 2017 Aug 17;17(1):106. doi: 10.1186/s12871-017-0401-8. PMID 28818054
- [Derived] Soltesz S, Stark C, Noe KG, Anapolski M, Mencke T. Monitoring recovery from rocuronium-induced neuromuscular block using acceleromyography at the trapezius versus the adductor pollicis muscle: an observational trial. Can J Anaesth. 2016 Jun;63(6):709-17. doi: 10.1007/s12630-016-0609-y. Epub 2016 Feb 10. PMID 26864194